CLINICAL TRIAL: NCT06071195
Title: All-in-One Prostate Cancer Staging with MRI
Acronym: AllinOne_MRI
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Collaborators: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other); Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 1537
Record Dates: First submitted 2023-10-03; First posted 2023-10-06 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Staging; Whole-Body Magnetic Resonance Imaging
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Prostate Cancer Patients: Patients will undergo a combined whole-body MRI + multiparametric prostate MRI examination along with routine staging examinations (PET, CT / bone scintigraphy).
  Reporting will be performed without and with reference to the whole-body MRI examination. Differences in the resulting staging and in management recommendations based on the two reportings will be recorded.
  Interventions: Diagnostic Test: Prostate Cancer Patients

INTERVENTIONS:
Diagnostic Test: Prostate Cancer Patients — see arm/group description

SUMMARY:
Prior to treatment, it is essential to assess not only the extent of prostate cancer within the prostate, but also to determine whether the disease has initiated metastatic spread. Whole-body MRI has become a viable option for the detection of metastatic disease derived from a number of cancers, but is typically performed in a separate scanning session to an initial dedicated prostate MRI in which the local disease is assessed. In patients known to be at high risk for significant prostate cancer prior to this initial MRI, and thus highly likely to proceed to treatment, this delays arriving at a definitive treatment decision. The investigators will evaluate the sensitivity of a protocol that combines bi-parametric prostate MRI, performed according to PI-RADS v2.1 guidelines, with a whole-body MRI based on the METastasis Reporting and Data System for Prostate Cancer (MET-RADS-P) guidelines, for an All-in-One, local and systemic staging of intermediate-favorable or high risk prostate cancer patients. The resulting staging decisions will be compared to the results of systemic staging with those obtained by computed tomography and bone scintigraphy in the standard staging pathway.

DETAILED DESCRIPTION:
Accurate tumor staging for unfavorable intermediate- and high-risk prostate cancer patients should underpin both prognostication and management decisions. This void necessitates evaluation of the local, primary disease as well as spread to distant sites including lymph nodes and possible distant metastases.

Multi-parametric magnetic resonance imaging (mp-MRI) has become the reference standard practice for local imaging-based assessment in prostate cancer (PCa). Whole-body MRI (WB-MRI) is seeing growing for detection of distant, metastatic disease, and is particularly suited to detection of bone metastases, which are common in PCa. The possibility of a one-stop staging modality has been raised, wherein mp-MRI + whole body MRI (WB-MRI) would be used to further assess nodal and metastatic disease status in a single sitting. Currently however, international guidelines consider bone scintigraphy (BS) and pelvic computed tomography (CT) for distant disease to be the mainstays of imaging-based staging decisions. A further concern with transitioning to All-in-One prostate staging with MRI relates to the duration of scanning required, as an excessive scan duration is likely to lead to patient discomfort, motion and consequently reduce image quality.

The prostate imaging reporting and data system (PI-RADS) v2.1 standard published by Turkbey et al. provides guidelines for mp-MRI of the prostate that are widely used as the basis for assessment of local, primary PCa. Recent evidence suggests that some components of the PI-RADS mp-MRI protocol are of little or no benefit to men with a very high risk of aggressive PCa, defined as prostate specific antigen (PSA) ≥10 ng/mL and + digital rectal exam, even before initial biopsy or repeated biopsy. In particular, dynamic contrast enhanced (DCE) imaging and T2-weighted images (T2WI) in a third orthogonal plane does not improve the overall accuracy of mp-MRI. Therefore, biparametric MRI (bp-MRI; i.e. T2WI in two planes, diffusion-weighted imaging (DWI, without contrast agent injection)) has been suggested to reduce examination time and cost, while retaining sufficient diagnostic accuracy to "rule out" high-grade PCa in biopsy-naïve men.

WB-MRI offers greater sensitivity and diagnostic accuracy for bone and nodal disease than BS and conventional CT. Further, a meta-analysis by Woo et al. has shown MRI (DWI + conventional sequences) to have excellent sensitivity and specificity in particular for detection of bone metastases in patients with PCa. The pooled per-patient sensitivity and specificity of MRI in the 10 studies included in the meta-analysis were 0.96 (95% confidence interval (CI) 0.87-0.99) and 0.98 (95% CI 0.93-0.99), respectively. Similar performance for WB-MRI is reported in the meta-analysis of Shen et al. who found the diagnostic performance of WB-MRI to be similar to that of choline PET/CT, with both being superior to BS in the detection of bone metastases. The pooled sensitivities and specificities in this meta-analysis were 0.97/0.95 and 0.79/0.82 for WB-MRI and BS respectively. WB-MRI appears to be more accurate than conventional CT, which not surprising the pooled sensitivities and specificities of CT alone have been reported as 0.42 and 0.82 in a pair of meta-analyses . A recent work by Johnston et al., found that a WB-MRI protocol consisting of unenhanced T1-weighted DIXON and diffusion-weighted scans provides much higher diagnostic accuracy than BS (sensitivity/specificity 0.90/0.88 vs 0.60/1.00) for the primary staging of intermediate- and high-risk PCa. They also found high and very similar sensitivities/specificities for WB-MRI and BS in respect to nodal disease, with values of 1.00/0.96 and 1.00/0.82 for N1 disease and 0.75/ 0.93 and 0.75/0.92 for M1a disease respectively.

The investigators are continuing their studies into the role and the added value of WB-MRI in oncologic patients with advanced cancer (prostate, breast, melanoma], lymphoma).

The investigators propose to evaluate the sensitivity of a protocol that combines bp-MRI of the prostate, following the PI-RADS v2.1 guideline, with WB-MRI based on MET-RADS-P guidelines, for an All-in-One, local and systemic staging of unfavorable intermediate- and high-risk prostate cancer patients and to compare the results of systemic staging with those obtained with CT and BS in the standard staging pathway. The combination of bp-MRI and WB-MRI is expected to require a scan time of roughly 40 minutes, allowing it to be performed in a conventional mp-MRI scan time allotment.

ELIGIBILITY:
Inclusion Criteria:

* at least one of: International Society of Urological Pathology Grade Group ≥ 3 (Gleason Score ≥ 4+3); cT3 initial diagnosis with any PSA level; PSA ≥ 20 ng/mL with any Gleason score;
* and all the following: Signed informed consent; Patients eligible to active treatment (either radical prostatectomy or radiotherapy) and/or hormone therapy; Life expectancy ≥ 10 years;

Exclusion Criteria:

* Contraindications to MRI (e.g. severe claustrophobia or MRI unsafe device);
* Previous or ongoing hormone therapy or radiation therapy for prostate cancer;
* Significant intercurrent morbidity that, in the judgment of the investigator, would limit compliance with study protocols;
* Previous mp-MRI performed within six weeks of the outpatient visit and compliant with PI-RADS v2.1 guidelines;
* Prostate cancer with significant sarcomatoid or spindle cell or neuroendocrine small cell components;

Min Age: 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: unfavorable intermediate- and high-risk prostate cancer patients
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2026-06-22 (Estimated); Study Completion 2026-08-22 (Estimated)

PRIMARY OUTCOMES:
Staging Sensitivity | 1 year
  Sensitivity (SE) of the evaluated diagnostic procedures based on the case report forms (CRFs) compiled at the time of reporting

SECONDARY OUTCOMES:
Staging Specificity | 1 year
  Specificity (SP) and the overall accuracy of the evaluated diagnostic procedures based on the CRFs compiled at the time of reporting

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Petralia, MD, Principal Investigator — European Institute of Oncology, IEO IRCCS
Locations (3):
- Italy (3):
  - Spedali Civili di Brescia, Brescia, BS
  - Istituto Europeo di Oncologia, Milan, MI
  - Azienda Ospedaliera Universitaria Integrata di Verona, Ospedale Borgo Roma, Verona, VR

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bjurlin MA, Rosenkrantz AB, Beltran LS, Raad RA, Taneja SS. Imaging and evaluation of patients with high-risk prostate cancer. Nat Rev Urol. 2015 Nov;12(11):617-28. doi: 10.1038/nrurol.2015.242. Epub 2015 Oct 20. PMID 26481576
- [Background] Turkbey B, Rosenkrantz AB, Haider MA, Padhani AR, Villeirs G, Macura KJ, Tempany CM, Choyke PL, Cornud F, Margolis DJ, Thoeny HC, Verma S, Barentsz J, Weinreb JC. Prostate Imaging Reporting and Data System Version 2.1: 2019 Update of Prostate Imaging Reporting and Data System Version 2. Eur Urol. 2019 Sep;76(3):340-351. doi: 10.1016/j.eururo.2019.02.033. Epub 2019 Mar 18. PMID 30898406
- [Background] Pasoglou V, Larbi A, Collette L, Annet L, Jamar F, Machiels JP, Michoux N, Vande Berg BC, Tombal B, Lecouvet FE. One-step TNM staging of high-risk prostate cancer using magnetic resonance imaging (MRI): toward an upfront simplified "all-in-one" imaging approach? Prostate. 2014 May;74(5):469-77. doi: 10.1002/pros.22764. Epub 2013 Dec 24. PMID 24375774
- [Background] Morote J, Celma A, Roche S, de Torres IM, Mast R, Semedey ME, Regis L, Planas J. Who Benefits from Multiparametric Magnetic Resonance Imaging After Suspicion of Prostate Cancer? Eur Urol Oncol. 2019 Nov;2(6):664-669. doi: 10.1016/j.euo.2018.11.009. Epub 2018 Dec 14. PMID 31411977
- [Background] Woo S, Suh CH, Kim SY, Cho JY, Kim SH, Moon MH. Head-to-Head Comparison Between Biparametric and Multiparametric MRI for the Diagnosis of Prostate Cancer: A Systematic Review and Meta-Analysis. AJR Am J Roentgenol. 2018 Nov;211(5):W226-W241. doi: 10.2214/AJR.18.19880. Epub 2018 Sep 21. PMID 30240296
- [Background] Choi MH, Kim CK, Lee YJ, Jung SE. Prebiopsy Biparametric MRI for Clinically Significant Prostate Cancer Detection With PI-RADS Version 2: A Multicenter Study. AJR Am J Roentgenol. 2019 Apr;212(4):839-846. doi: 10.2214/AJR.18.20498. Epub 2019 Feb 19. PMID 30779662
- [Background] Obmann VC, Pahwa S, Tabayayong W, Jiang Y, O'Connor G, Dastmalchian S, Lu J, Shah S, Herrmann KA, Paspulati R, MacLennan G, Ponsky L, Abouassaly R, Gulani V. Diagnostic Accuracy of a Rapid Biparametric MRI Protocol for Detection of Histologically Proven Prostate Cancer. Urology. 2018 Dec;122:133-138. doi: 10.1016/j.urology.2018.08.032. Epub 2018 Sep 7. PMID 30201301
- [Background] Boesen L, Norgaard N, Logager V, Balslev I, Bisbjerg R, Thestrup KC, Winther MD, Jakobsen H, Thomsen HS. Assessment of the Diagnostic Accuracy of Biparametric Magnetic Resonance Imaging for Prostate Cancer in Biopsy-Naive Men: The Biparametric MRI for Detection of Prostate Cancer (BIDOC) Study. JAMA Netw Open. 2018 Jun 1;1(2):e180219. doi: 10.1001/jamanetworkopen.2018.0219. PMID 30646066
- [Background] Niu XK, Chen XH, Chen ZF, Chen L, Li J, Peng T. Diagnostic Performance of Biparametric MRI for Detection of Prostate Cancer: A Systematic Review and Meta-Analysis. AJR Am J Roentgenol. 2018 Aug;211(2):369-378. doi: 10.2214/AJR.17.18946. Epub 2018 Jun 12. PMID 29894216
- [Background] Lecouvet FE, El Mouedden J, Collette L, Coche E, Danse E, Jamar F, Machiels JP, Vande Berg B, Omoumi P, Tombal B. Can whole-body magnetic resonance imaging with diffusion-weighted imaging replace Tc 99m bone scanning and computed tomography for single-step detection of metastases in patients with high-risk prostate cancer? Eur Urol. 2012 Jul;62(1):68-75. doi: 10.1016/j.eururo.2012.02.020. Epub 2012 Feb 17. PMID 22366187
- [Background] Woo S, Suh CH, Kim SY, Cho JY, Kim SH. Diagnostic Performance of Magnetic Resonance Imaging for the Detection of Bone Metastasis in Prostate Cancer: A Systematic Review and Meta-analysis. Eur Urol. 2018 Jan;73(1):81-91. doi: 10.1016/j.eururo.2017.03.042. Epub 2017 Apr 12. PMID 28412063
- [Background] Shen G, Deng H, Hu S, Jia Z. Comparison of choline-PET/CT, MRI, SPECT, and bone scintigraphy in the diagnosis of bone metastases in patients with prostate cancer: a meta-analysis. Skeletal Radiol. 2014 Nov;43(11):1503-13. doi: 10.1007/s00256-014-1903-9. Epub 2014 May 20. PMID 24841276
- [Background] Hovels AM, Heesakkers RA, Adang EM, Jager GJ, Strum S, Hoogeveen YL, Severens JL, Barentsz JO. The diagnostic accuracy of CT and MRI in the staging of pelvic lymph nodes in patients with prostate cancer: a meta-analysis. Clin Radiol. 2008 Apr;63(4):387-95. doi: 10.1016/j.crad.2007.05.022. Epub 2008 Feb 4. PMID 18325358
- [Background] Evangelista L, Guttilla A, Zattoni F, Muzzio PC, Zattoni F. Utility of choline positron emission tomography/computed tomography for lymph node involvement identification in intermediate- to high-risk prostate cancer: a systematic literature review and meta-analysis. Eur Urol. 2013 Jun;63(6):1040-8. doi: 10.1016/j.eururo.2012.09.039. Epub 2012 Sep 25. PMID 23036576
- [Background] Johnston EW, Latifoltojar A, Sidhu HS, Ramachandran N, Sokolska M, Bainbridge A, Moore C, Ahmed HU, Punwani S. Multiparametric whole-body 3.0-T MRI in newly diagnosed intermediate- and high-risk prostate cancer: diagnostic accuracy and interobserver agreement for nodal and metastatic staging. Eur Radiol. 2019 Jun;29(6):3159-3169. doi: 10.1007/s00330-018-5813-4. Epub 2018 Dec 5. PMID 30519933
- [Background] Padhani AR, Lecouvet FE, Tunariu N, Koh DM, De Keyzer F, Collins DJ, Sala E, Schlemmer HP, Petralia G, Vargas HA, Fanti S, Tombal HB, de Bono J. METastasis Reporting and Data System for Prostate Cancer: Practical Guidelines for Acquisition, Interpretation, and Reporting of Whole-body Magnetic Resonance Imaging-based Evaluations of Multiorgan Involvement in Advanced Prostate Cancer. Eur Urol. 2017 Jan;71(1):81-92. doi: 10.1016/j.eururo.2016.05.033. Epub 2016 Jun 14. PMID 27317091
- [Background] Pricolo P, Ancona E, Summers P, Abreu-Gomez J, Alessi S, Jereczek-Fossa BA, De Cobelli O, Nole F, Renne G, Bellomi M, Padhani AR, Petralia G. Whole-body magnetic resonance imaging (WB-MRI) reporting with the METastasis Reporting and Data System for Prostate Cancer (MET-RADS-P): inter-observer agreement between readers of different expertise levels. Cancer Imaging. 2020 Oct 27;20(1):77. doi: 10.1186/s40644-020-00350-x. PMID 33109268
- [Background] Zugni F, Ruju F, Pricolo P, Alessi S, Iorfida M, Colleoni MA, Bellomi M, Petralia G. The added value of whole-body magnetic resonance imaging in the management of patients with advanced breast cancer. PLoS One. 2018 Oct 12;13(10):e0205251. doi: 10.1371/journal.pone.0205251. eCollection 2018. PMID 30312335
- [Background] Petralia G, Padhani A, Summers P, Alessi S, Raimondi S, Testori A, Bellomi M. Whole-body diffusion-weighted imaging: is it all we need for detecting metastases in melanoma patients? Eur Radiol. 2013 Dec;23(12):3466-76. doi: 10.1007/s00330-013-2968-x. Epub 2013 Jul 25. PMID 23884300
- [Background] Montoro J, Laszlo D, Zing NP, Petralia G, Conte G, Colandrea M, Martinelli G, Preda L. Comparison of whole-body diffusion-weighted magnetic resonance and FDG-PET/CT in the assessment of Hodgkin's lymphoma for staging and treatment response. Ecancermedicalscience. 2014 May 15;8:429. doi: 10.3332/ecancer.2014.429. eCollection 2014. PMID 24963346